CLINICAL TRIAL: NCT02902094
Title: Improving Outcomes in Fistula Intervention: A Prospective, Patient Blinded, Phase 3, Randomised Controlled Trial of Drug Eluting Balloons in the Angioplasty of Native Haemodialysis Access Arteriovenous Fistula Outflow Stenosis (DeVA)
Brief Title: Drug Eluting Balloon Venoplasty in AV Fistula Stenosis
Acronym: DeVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRK5479
Record Dates: First submitted 2016-06-21; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Native Arteriovenous Fistula; Stenosis
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Drug eluting angioplasty balloons
  Interventions: Device: Drug eluting balloons
- Control (Active Comparator): Non-drug eluting balloons
  Interventions: Device: Non drug eluting balloons

INTERVENTIONS:
Device: Drug eluting balloons
  Arms: Experimental
Device: Non drug eluting balloons
  Arms: Control

SUMMARY:
DeVA is a single blinded, prospective, multicentre RCT designed to determine the safety and effectiveness of a drug eluting angioplasty balloon compared with a standard angioplasty balloon in patients with symptomatic native AV fistula stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Arteriovenous (AV) fistulas with stenosis requiring percutaneous angioplasty identified on routine diagnostic imaging or causing clinical concern on dialysis.
* Fistula has been in use for at least 1 month and is > 6 weeks old
* Brachiocephalic AV fistula
* Brachiobasilic AV fistula
* Radiocephalic AV fistula (both proximal and distal)
* Participant >/=18 yrs old
* Index lesion is less then the length of the DEB, and the reference vessel diameter is appropriate for treatment with the size range of DEB (4mm - 8mm diameter)
* Participant is able to give valid informed consent

Exclusion Criteria:

* Allergy to iodinated Intravenous contrast
* Allergy to Paclitaxel
* Prosthetic grafts
* Long or tandem lesions that cannot be treated with a single DEB
* Thrombosed Arterio-Venous fistulas
* Women who are breastfeeding, pregnant or intending to become pregnant
* Participants of child-bearing age who are unwilling to use a reliable form of contraception for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Patency | 12 months
  Primary end point is a composite of one or more of :
  * >50% stenosis of index lesion requiring re-intervention
  * Re-intervention of index lesion due to clinical indications without 50% re-stenosis
  * Fistula failure

SECONDARY OUTCOMES:
Technical success | Time of baseline index intervention
  Defined as <30% residual stenosis using only the study balloon to which the patient was randomised
Assisted technical success of balloon angioplasty | At time of baseline index intervention
  Defined as <30% residual stenosis using adjunctive procedures in addition to study balloon
Successful use of fistula for dialysis | In the 12 months following baseline index intervention
  Defined as successful use of the fistula for dialysis using 2 needles on at least one occasion
Secondary patency of the access circuit | In the 12 months following baseline index intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, Dr, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No